CLINICAL TRIAL: NCT00407914
Title: A Double-Masked, Randomized, Multi-Center, 2-Arm Parallel Study Comparing the Safety and Effectiveness of Aquamid and Restylane for the Aesthetic Treatment of Nasolabial Folds
Brief Title: Safety and Effectiveness of Aquamid as Compared to Restylane for the Aesthetic Treatment of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contura (Industry)
Responsible Party: Silvia G Codony, Clinical Research Director, Contura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONAQ-US01
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Facial Wrinkles
Keywords: wrinkles; soft tissue filler; Aquamid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Aquamid
  Interventions: Device: Aquamid
- 2 (Active Comparator): Restylane
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Aquamid — Subcutaneous injection
  Arms: 1
Device: Restylane — Injection in dermis
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of Aquamid and Restylane in aesthetically enhancing nasolabial folds 6 months after treatment and to evaluate the safety of Aquamid through 12 months after treatment.

The study includes an extended follow up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* interested on soft tissue augmentation for the nasolabial folds
* moderate to severe nasolabial fold

Exclusion Criteria:

* sensitivity to anesthetics
* allergy to hyaluronic acid
* previous treatment with permanent fillers in the treated area
* recent previous aesthetic procedure in the treatment area
* infected skin areas or autoimmune diseases affecting the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Wrinkle Assessment Scale | Baseline, 3, 6, 9, 12 Months
Adverse device effects | continuosly

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale | Optimal treatment, 3, 6, 9 and 12 Months
Injection site reactions | After injection
Adverse events | continuosly

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Codony, Study Director — Contura
Locations (1):
- White Plains, New York, United States

REFERENCES:
- [Background] von Buelow S, von Heimburg D, Pallua N. Efficacy and safety of polyacrylamide hydrogel for facial soft-tissue augmentation. Plast Reconstr Surg. 2005 Sep 15;116(4):1137-46; discussion 1147-8. doi: 10.1097/01.prs.0000179349.14392.a4. PMID 16163108